CLINICAL TRIAL: NCT06270030
Title: A Single-Center, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of LNZ101 and LNZ100 Ophthalmic Solutions in Chinese Healthy Adult Subjects With Presbyopia
Brief Title: Safety, Tolerability and Pharmacokinetics of LNZ101 and LNZ100 Ophthalmic Solutions in Healthy Adult Chinese With Presbyopia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corxel Pharmaceuticals (Industry)
Collaborators: LENZ Therapeutics, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JX07002; CTR20240460 (Other: China Center for Drug Evaluation (CDE), NMPA)
Record Dates: First submitted 2024-02-06; First posted 2024-02-21 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Presbyopia
Keywords: Presbyopia; LNZ100; LNZ101
MeSH Terms: conditions — Presbyopia | interventions — aceclidine; Brimonidine Tartrate; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LNZ101 (Aceclidine /Brimonidine) ophthalmic solution (Experimental): Drug: Aceclidine/Brimonidine ophthalmic solution Other Names: LNZ101
  Interventions: Drug: LNZ101 (Aceclidine /Brimonidine) ophthalmic solution
- LNZ100 (Aceclidine) ophthalmic solution (Experimental): Drug: Aceclidine ophthalmic solution Other Names: LNZ100
  Interventions: Drug: LNZ100 (Aceclidine) ophthalmic solution
- Placebo (Vehicle) ophthalmic solution (Placebo Comparator): Drug: Placebo (Vehicle) ophthalmic solution Other Names: NA
  Interventions: Drug: Placebo (Vehicle) ophthalmic solution

INTERVENTIONS:
Drug: LNZ101 (Aceclidine /Brimonidine) ophthalmic solution — Once daily from day 1 to day 8; Everyday, subject will be administered with 1 drop in each eye followed by another drop in each eye 2 minutes later
  Arms: LNZ101 (Aceclidine /Brimonidine) ophthalmic solution
Drug: LNZ100 (Aceclidine) ophthalmic solution — Once daily from day 1 to day 8; Everyday, subject will be administered with 1 drop in each eye followed by another drop in each eye 2 minutes later
  Arms: LNZ100 (Aceclidine) ophthalmic solution
Drug: Placebo (Vehicle) ophthalmic solution — Once daily from day 1 to day 8; Everyday, subject will be administered with 1 drop in each eye followed by another drop in each eye 2 minutes later
  Arms: Placebo (Vehicle) ophthalmic solution

SUMMARY:
Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of LNZ101 and LNZ100 Ophthalmic Solutions in Chinese Healthy Adult Subjects with Presbyopia

DETAILED DESCRIPTION:
A Single-Center, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of LNZ101 and LNZ100 Ophthalmic Solutions in Chinese Healthy Adult Subjects with Presbyopia

ELIGIBILITY:
Inclusion Criteria

1. Be able and willing to provide written informed consent prior to any study procedure being performed.
2. Be able to and willing to use investigational products per study requirements and attend all study assessments, including admission to and stay in the CRU on required study days.
3. Be Chinese healthy male or female subjects aged 45-75 years (inclusive) at screening.
4. Be diagnosed and documented to have presbyopia by the investigator at the screening visit.

Exclusion Criteria:

1. Have known contraindications or sensitivity to the use of any of the investigational products or its components, or any other medications required by the protocol.
2. Have any active systemic or ocular disorder that has a potential risk to or impact on subject safety, study process or study results other than refractive disorder.
3. Have presence of any abnormality of the lids, ocular surface, or lacrimal duct system that in the investigator's opinion could affect ophthalmic solution absorption in either eye.
4. Have prior (within 14 days of the first dose), current or anticipated use of any contact lenses during study participation.
5. Be ineligible for this trial in the opinion of the investigator.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 1 and Day 8
  Maximum plasma concentrations of LNZ100 and LNZ101
Tmax | Day 1 and Day 8
  Time of maximum plasma concentrations of LNZ100 and LNZ101
AUC0-t | Day 1 and Day 8
  Area under the concentration-time curve from time 0 to time t of LNZ100 and LNZ100
AUC0-∞ | Day 1 and Day 8
  Area under the concentration-time curve from time 0 to infinity of LNZ100 and LNZ101
T1/2 | Day 1 and Day 8
  Terminal half-life of LNZ100 and LNZ101
Safety: adverse event reporting | up to 23 days
  The number of patients who experience one or more AE during the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Larry Li, Doctor, Study Director — Corxel Pharmaceuticals
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China